CLINICAL TRIAL: NCT03715166
Title: A 6-month Randomised, Double-blind, Placebo Controlled Multicentre Parallel Group Study to Evaluate Efficacy and Safety of Bumetanide 0.5mg Twice a Day Followed by an Open Label Active 6-month Treatment Period With Bumetanide (0.5mg Twice a Day) and a 6 Weeks Discontinuation Period After Treatment Stop.
Brief Title: Efficacy and Safety of Bumetanide Oral Liquid Formulation in Children and Adolescents Aged From 7 to Less Than 18 Years Old With Autism Spectrum Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The 6-month efficacy analysis did not show any significant difference between bumetanide versus placebo in the treatment of ASD in the overall studied population. No unexpected safety concerns were identified.
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-95008-001; 2017-004419-38 (EudraCT Number)
Record Dates: First submitted 2018-10-12; First posted 2018-10-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Bumetanide

STUDY DESIGN:
Intervention Model Description: 6-month, randomized, double-blind, placebo-controlled, parallel groups followed by an open label active 6-month treatment period with bumetanide.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bumetanide/S95008 (Experimental)
  Interventions: Drug: Bumetanide Oral Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide Oral Solution — Oral Solution dosed at 0.5mg/mL Taken twice daily
  Arms: Bumetanide/S95008
Drug: Placebo — Oral Solution Taken twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and the safety of bumetanide/S95008 in the improvement of Autism Spectrum Disorder core symptoms.

DETAILED DESCRIPTION:
The present study (CL3-95008-001) was performed in children and adolescents from 7 to less than 18 years old presenting with ASD. A 6-month double-blind treatment period was performed in which efficacy and safety of bumetanide 0.5mg BID were assessed versus placebo. This double-blind period was followed by a 6-month open label treatment period of bumetanide 0.5mg BID in which long term safety was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 7 to less than 18 years
* Out patients
* Primary diagnosis of ASD as per Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria
* Criteria met for ASD on Autism Diagnostic Observation Schedule (ADOS-2) and Autism Diagnosis Interview Revised (ADI-R)
* CGI (Clinical Global Impression) - Severity rating Score ≥ 4
* Childhood Autism Rating Scale second edition (CARS2-ST or HF) total raw score ≥ 34
* Social responsiveness Scale second edition total score (SRS-2 T-Score) ≥ 66
* Absence of known monogenic syndrome (Fragile X, Rett syndrome ...)
* Absence of any clinically significant abnormality likely to interfere with the conduct of the study according to the judgment of the investigator

Exclusion Criteria:

* Patients not able to follow the study assessments defined by the protocol, with the exception of self-rating questionnaires which will be assessed by parent/legal representative/caregiver for those patients unable to complete them
* Patients having a high suicidal risk according to the investigator judgement
* Chronic renal dysfunction
* Chronic cardiac dysfunction
* Patient with unstable psychotherapy, behavioural, cognitive or cognitive-behavioural therapy
* Severe electrolyte imbalance that is likely to interfere with the study conduct or evaluation

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale, Second Edition (CARS2) total raw score | Change from baseline to 6 month
  Efficacy criterion The CARS2 is a 15 item rated instrument. The rating values given for the 15 areas are summed to produce a Total score.

SECONDARY OUTCOMES:
Social Responsiveness Scale, Second Edition (SRS-2) total raw score | Change from baseline to 6 month
  Efficacy criterion 65 items scale measuring symptoms associated with autism
Clinical Global Impression - Global Improvement (CGI-I) score | At 6 months
  Efficacy criterion Scale which assesses the severity of the illness and the global improvement of the patient under study treatment
Vineland Adaptative Behaviour Sales, Second Edition (VABS II) subscores | Change from baseline to 6 month
  Efficacy criterion Scale designated to measure adaptative behaviour
Adverse events and Paediatric Adverse Event Rating Scale (PAERS) | On average of 52 weeks
  Safety criterion Inventory report used to identify signs/symptoms experienced by the patient since the study treatment initiation.
Abnormalities in 12-leads electrocardiogram (ECG) parameters | selection visit/Week004/Week008/Week012/Week 026/Week030/Week034/Week038/Week052
  Safety criterion
Renal ultrasound | selection visit/Week026/Week052
  Safety criterion Assessment of the renal function
the Columbia Suicide Severity Rating Scale Children's version (C-SSRS-C) | Week000/Week012/Week026/Week038/Week052
  Scale which assesses suicidal ideation and suicidal behaviour
Tanner stage | Week000/Week026/Week052
  Safety criterion Assessment of Pubertal development
Acceptability and palatability questionnaire | Week026
  Acceptability and palatability criterion Assessment of the ease of use to use the dosing device
Paediatric Quality of Life Inventory (PedsQL) questionnaire | Week000/Week004/Week012/Week026/Week030/Week038/Week052
  Quality of Life criterion Assessment of parent/legal representative perception of patient health related quality of life

CONTACTS AND LOCATIONS:
Locations (45):
- Brazil (5):
  - Trial Tech em Pesquisas com Medicamentos Ltda, Curitiba
  - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza
  - Hospital São Vicente de Paulo, Passo Fundo
  - Universidade Federal de São Paulo, Escola Paulista de Medicina, São Paulo
  - Faculdade de Medicina da Universidade de São Paulo - Departamento de Psiquiatria, São Paulo
- France (9):
  - GSC CHU-LENVAL Centre ressource autisme, Nice, Alpes-Maritimes
  - Centre d'Investigation Clinique de Lyon, Bron, Auvergne-Rhône-Alpes
  - Hôpital Le Vinatier CRA Rhône-Alpes, Bat 211, Bron, Auvergne-Rhône-Alpes
  - Hôpitaux Universitaires de Strasbourg Service de Psychiatrie de l'Enfant et de l'Adolescent, Strasbourg, Grand Est
  - Hôpital Robert Debré Service de Psychiatrie de l'enfant et de l'adolescent, Paris, Il de France
  - CHU Rouen, Rouen, Normandy
  - Centre Hospitalier du Rouvray Centre de Ressources pour l'Autisme, Sotteville-lès-Rouen, Normandy
  - Centre Hospitalier Charles Perrens CRA Aquitaine, Bordeaux, Nouvelle-Aquitaine
  - Hôpital des Enfants-Pellegrin, Bordeaux, Nouvelle-Aquitaine
- Germany (3):
  - Universitätsklinikum Freiburg, Zentrum für Psychische Erkrankungen, Klinik für Psychiatrie, Psychotherapie und Psychosomatik im Kindes- und Jugendalter, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinik für Psychiatrie und Psychotherapie des Kindes- und Jugendalters am Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Klinik und Poliklinik für Kinder- und Jugendpsychiatrie und, Dresden, Saxony (Sachsen)
- Hungary (4):
  - Vadaskert Korhaz es Szakambulancia, Budapest
  - Servus Salvus Kft., Budapest
  - Bekes Megyei Kozponti Korhaz Gyermek es ifjusagpszichiatriai osztaly, Gyula
  - Szegedi Tudományegyetem Szent-Gyorgy Albert Klinikai Kozpont Gyermekgyógyászati Klinika Gyermek es Ifjusagpszichiátriai o, Szeged
- Italy (7):
  - Unità Semplice di Psichiatria Infantile Policlinico Universitario di Napoli - Università Federico II, Napoli, Campania
  - Neuro Riabilitazione/Psicopatologia dell'età evolutiva Istituto Scientifico Medea - Bosisio Parini, Bosisio Parini, Lombardy
  - U.O. di Neuropsichiatria Infantile Fondazione Istituto Neurologico Nazionale Casimiro Mondino Istituto di Ricovero e Cura a Carattere Scientifico, Pavia, Lombardy
  - Clinica di Neuropsichiatria dell'Infanzia e dell'Adolescenza Ospedale Pediatrico-Microcitemico, Cagliari, Sardinia
  - Programma Interdipartimentale "Autismo 0-90" A.O.U. Policlinico "Gaetano Martino", Messina, Sicily
  - U.O.C. Psichiatria dello Sviluppo IRCCS Fondazione Stella Maris, Calambrone, Tuscany
  - U.O. di Neuropsichiatria Infantile Azienda Ospedaliera Universitaria Senese, Siena, Tuscany
- Accare Groningen, Groningen, Netherlands
- Poland (5):
  - Samodzielny Publiczny Dziecięcy Szpital Kliniczny w Warszawie Oddział Kliniczny Psychiatrii Wieku Rozwojowego, Warsaw, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej Gdańskie Centrum Zdrowia Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Badań Klinicznych PI-House sp. z o.o, Gdansk
  - Fundacja SYNAPSIS ul., Warsaw
  - NAVICULA Centrum Diagnozy i Terapii Autyzmu w Łodzi, Lodz, Łódź Voivodeship
- Centro Hospitalar e Universitario de Coimbra Hospital Pediatrico, Coimbra, Portugal
- Spain (7):
  - Hospita Mutua de Terrassa, Terrassa, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Niño Jesus, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
- United Kingdom (3):
  - Forward Thinking Birmingham_Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - ReCognition Health, London
  - The Winnicott Centre, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Fuentes J, Parellada M, Georgoula C, Oliveira G, Marret S, Crutel V, Albarran C, Lambert E, Penelaud PF, Ravel D, Ben Ari Y. Bumetanide oral solution for the treatment of children and adolescents with autism spectrum disorder: Results from two randomized phase III studies. Autism Res. 2023 Oct;16(10):2021-2034. doi: 10.1002/aur.3005. Epub 2023 Oct 4. PMID 37794745
- [Derived] Hawken N, Falissard B, Choquet C, Francois C, Tardu J, Schmid R. Exit interviews from two randomised placebo-controlled phase 3 studies with caregivers of young children with autism spectrum disorder. Front Child Adolesc Psychiatry. 2024 Jun 5;3:1236340. doi: 10.3389/frcha.2024.1236340. eCollection 2024. PMID 39816573
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/